CLINICAL TRIAL: NCT01107899
Title: Recovery of Platelet Function After a Loading Dose of Prasugrel or Clopidogrel in Aspirin-Treated Subjects Presenting With Symptoms of Acute Coronary Syndromes
Brief Title: Study to Learn When Platelets Return to Normal After One Loading Dose of Anti-platelet Drugs in Patients With Symptoms of Acute Coronary Syndromes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to Enrollment futility
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11983; H7T-MC-TACM (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Results first posted 2012-01-12 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes; Angina; Platelet Function; Coronary Angiography; Clinical Symptoms of Angina; Positive Stress Test
MeSH Terms: conditions — Acute Coronary Syndrome; Angina Pectoris | interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- clopidogrel 600 mg (Active Comparator)
  Interventions: Drug: clopidogrel
- prasugrel 60 mg (Active Comparator)
  Interventions: Drug: prasugrel
- prasugrel 30 mg (Experimental)
  Interventions: Drug: prasugrel

INTERVENTIONS:
Drug: clopidogrel — taken orally, day one, single dose
  Arms: clopidogrel 600 mg
Drug: prasugrel — taken orally, day one, single dose
  Other Names: Efient®; Effient®; LY640315; CS747
  Arms: prasugrel 30 mg; prasugrel 60 mg

SUMMARY:
To investigate how platelets recover to normal function in subjects who have symptoms of a heart attack or unstable angina and who get a loading dose of prasugrel or clopidogrel for planned coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 to <80 years of age who present with any one of the following:
* symptoms of Acute Coronary Syndromes (ACS)
* clinical symptoms of angina, or a positive stress test or who return for routine follow up angiography post stent placement in whom co-administration of aspirin and a thienopyridine (that is, clopidogrel, ticlopidine, or prasugrel) is not contraindicated

Exclusion Criteria:

* Those presenting with ST-elevation MI (STEMI)
* histories of refractory ventricular arrhythmias
* an implanted defibrillator device
* congestive heart failure (NYHA Class III or above) within 6 months prior to screening
* significant hypertension
* subjects with a history or clinical suspicion of cerebral vascular malformations, transient ischaemic attack, or stroke
* bleeding disorders
* women known to be pregnant, who have given birth within the past 90 days, or who are breastfeeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich, Germany

REFERENCES:
- [Derived] Bernlochner I, Morath T, Brown PB, Zhou C, Baker BA, Gupta N, Jakubowski JA, Winters KJ, Schomig A, Kastrati A, Sibbing D. A prospective randomized trial comparing the recovery of platelet function after loading dose administration of prasugrel or clopidogrel. Platelets. 2013;24(1):15-25. doi: 10.3109/09537104.2011.654003. Epub 2012 Feb 28. PMID 22372531

RESULTS

PARTICIPANT FLOW:
Groups:
- Clopidogrel 600 mg: Clopidogrel 600 mg taken orally, day one, single dose (Loading Dose [LD])
- Prasugrel 60 mg: Prasugrel 60 mg taken orally, day one, single dose (Loading Dose [LD])
- Prasugrel 30 mg: Prasugrel 30 mg taken orally, day one, single dose (Loading Dose [LD])
Period: Overall Study
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Started | 10 | 10 | 9
Received at Least One Dose of Study Drug | 10 | 10 | 8
Loading Dose (LD) Intent to Treat (ITT) | 5 (Received LD and had evaluable pharmacodynamic (PD) measurements 24-hours post-LD.) | 10 (Received LD and had evaluable pharmacodynamic (PD) measurements 24-hours post-LD.) | 6 (Received LD and had evaluable pharmacodynamic (PD) measurements 24-hours post-LD.)
ITT Washout Population | 5 (ITT Washout Population (WP): Received LD, had evaluable baseline PD data (pre-LD) and post-LD.) | 10 (ITT Washout Population (WP): Received LD, had evaluable baseline PD data (pre-LD) and post-LD.) | 6 (ITT Washout Population (WP): Received LD, had evaluable baseline PD data (pre-LD) and post-LD.)
Primary Washout Population | 5 (Primary WP: Completed study with no missed visits, had evaluable PD data through Day 11.) | 10 (Primary WP: Completed study with no missed visits, had evaluable PD data through Day 11.) | 4 (Primary WP: Completed study with no missed visits, had evaluable PD data through Day 11.)
Completed | 5 | 10 | 5
Not Completed | 5 | 0 | 4
Not completed — Physician Decision | 5 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg | Total
Number analyzed (Participants) | 10 | 10 | 9 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 66.9 (8.54) | 65.6 (6.56) | 61.5 (10.01) | 64.8 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 9 | 8 | 7 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White | 10 | 10 | 9 | 29
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 10 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Returning to Baseline Platelet Function
Description: Participants were classified as having platelet function return to baseline after loading dose (LD) on the first day that P2Y12 Reaction Units (PRU) was no more than 60 PRU below baseline and remained in this range. PRU was assessed by Accumetrics Verify Now™ P2Y12. PRU represents the rate and extent of adenosine diphosphate (ADP)-stimulated platelet aggregation.
Time Frame: Days 3, 5, 7, 9, and 11
Population: Primary Washout Population: Included participants who completed the study, had evaluable pharmacodynamic (PD) data through Day 11. Participants with a missed visit were not included in the Primary Washout Population.
Measure: Number; unit: percentage of participants
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 5 | 10 | 4
percentage of participants
  Day 3 | 60.0 | 0 | 0
  Day 5 | 80.0 | 10.0 | 0
  Day 7 | 100.0 | 60.0 | 100.0
  Day 9 | 100.0 | 100.0 | 100.0
  Day 11 | 100.0 | 100.0 | 100.0

2. Secondary Outcome: The Day on Which 50%, 75% and 90% of Subjects Return to Baseline Platelet Function Following a Single LD of 30-mg or 60-mg Prasugrel or 600-mg Clopidogrel
Description: This outcome measure was not analyzed due to the limited sample size.
Time Frame: Up through 11 days
Population: Since this outcome measure was not analyzed due to the limited sample size, zero participants were included in the analysis.
Measure: Number; unit: days
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: The Day When the Proportion of Participants Who Return to Baseline Platelet Function in the 30-mg and 60-mg Prasugrel Groups is Similar to the 600-mg Clopidogrel Group at Day 5 and Day 7
Description: The day at which the proportion of participants who return to baseline platelet P2Y12 receptor function in the prasugrel 30 mg and 60 mg LD groups is similar (within 10% absolute difference) to the proportion of subjects who return to baseline platelet P2Y12 receptor function at day 5 and day 7 in the clopidogrel 600 mg LD group, obtained from Kaplan Meier curves for the primary washout population, was to be presented. This outcome measure was not analyzed due to the limited sample size.
Time Frame: Up through 11 days
Population: as for outcome 2
Measure: Number; unit: day
Arm/Group | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Days to the Return of Baseline Platelet Function Following One Loading Dose (LD)
Description: The return of baseline platelet function following one LD of prasugrel (30 mg or 60 mg) or 600 mg LD of clopidogrel assessed by Verify Now™ P2Y12 Reaction Units (VN-PRU). This outcome measure was not analyzed because it was not appropriate to estimate the days based on the non-inferiority approach due to the limited sample size.
Time Frame: Up through 11 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Effect of Initial Inhibition of Platelet Aggregation on the Day to Return to Baseline Platelet Function: VN-PRU
Description: To show effect of initial inhibition of platelet aggregation as measured by Accumetrics Verify Now™ P2Y12 on the day to return to baseline platelet function, a regression model was fitted with day to return as outcome variable and initial inhibition as fixed effect. Results are reported as the predicted day to return to baseline platelet function by derived VN-PRU percent (%) inhibition at 24 hours post LD. The derived VN-PRU % inhibition is calculated as a percent decrease of PRU from baseline using the following formula: ([PRU at baseline - PRU at 24 hours post LD]/PRU at baseline) x 100%.
Time Frame: Up through 11 days
Population: ITT Washout Population: All randomized participants who received study drug LD, had an evaluable baseline PD measurement (pre-LD), and had at least 1 evaluable PD measurement post-LD. One participant discontinued on Day 3 without returning to baseline and is not included in analysis.
Measure: Number; unit: days
Groups:
- All Treatments: Clopidogrel 600 mg taken orally, day one, single dose Prasugrel 30 and 60 mg taken orally, day one, single dose
  All treatments were combined into one group.
Arm/Group | All Treatments
Number analyzed (Participants) | 20
days
  20% Initial Inhibition | 3.2
  40% Initial Inhibition | 4.6
  60% Initial Inhibition | 6.0
  80% Initial Inhibition | 7.4
Statistical Analysis 1: Comparison: All Treatments; Test type: Superiority or Other; p < 0.001, Regression, Linear — P-value is for the overall effect of initial inhibition on the day to return to baseline platelet function

6. Secondary Outcome: Mean Number of Days to the Return of Baseline Platelet Function in All Treatment Arms (Adjusted for Level of Inhibition 24 Hrs Post-LD) by VN-PRU
Description: PRU was assessed by Accumetrics Verify Now™ P2Y12. PRU represents the rate and extent of adenosine diphosphate (ADP)-stimulated platelet aggregation. This outcome measure was not analyzed due to the limited sample size.
Time Frame: Up through 11 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Platelet Function 24 Hours Post Loading Dose
Description: PRU was assessed by Accumetrics Verify Now™ P2Y12. PRU represents the rate and extent of ADP-stimulated platelet aggregation.
Time Frame: 24 hours post-loading dose
Population: LD ITT population: All randomized participants who received an LD with evaluable PD measurements 24 hours post-LD.
Measure: Mean (Standard Deviation); unit: P2Y12 Reaction Units (PRU)
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 5 | 10 | 6
P2Y12 Reaction Units (PRU) | 193.0 (83.58) | 32.5 (20.79) | 70.0 (56.23)
Statistical Analysis 1: Comparison: Clopidogrel 600 mg vs Prasugrel 60 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; p-value was obtained from an analysis of covariance model with treatment as a fixed effect and the baseline value as a covariate
Statistical Analysis 2: Comparison: Clopidogrel 600 mg vs Prasugrel 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Prasugrel 60 mg vs Prasugrel 30 mg; Test type: Superiority or Other; p = 0.025, ANCOVA; [statistical method as in outcome 7, analysis 1]

8. Secondary Outcome: Percentage of Poor Pharmacodynamic Responders by Platelet Aggregation at 24 Hours Post-LD
Description: Platelet aggregation was assessed by Accumetrics Verify Now™ P2Y12, and poor responders were those with PRU greater than or equal to 230.
Time Frame: 24 hours post-loading dose
Population: LD ITT Population: All randomized participants who received an LD with evaluable PD measurements.
Measure: Number; unit: percentage of participants
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 5 | 10 | 6
percentage of participants | 40.0 | 0 | 0

9. Secondary Outcome: Extent of Initial Inhibition of Platelet Aggregation on the Return of Baseline Platelet Function: Light Transmission Aggregometry (LTA)
Description: Initial inhibition of platelet aggregation was measured by LTA at 5 and 20 μM ADP. Maximum platelet aggregation (MPA) is reported by day.
Time Frame: Up through 11 days
Population: ITT Washout Population: All randomized participants who received the study drug LD, had an evaluable baseline PD measurement (pre-LD), and had at least 1 evaluable PD measurement post-LD.
Measure: Mean (90% Confidence Interval); unit: percent platelet aggregation
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 5 | 10 | 6
percent platelet aggregation
  Baseline (20 μM ADP) (n=5, n=10, n=6) | 68.00 [61.82 to 74.18] | 72.70 [65.31 to 80.09] | 76.33 [66.76 to 85.91]
  Day 1 (20 μM ADP) (n=5, n=10, n=6) | 52.60 [32.96 to 72.24] | 27.30 [21.00 to 33.60] | 31.67 [22.51 to 40.82]
  Day 3 (20 μM ADP) (n=5, n=10, n=6) | 56.00 [40.25 to 71.75] | 42.50 [37.69 to 47.31] | 46.33 [33.38 to 59.28]
  Day 5 (20 μM ADP) (n=5, n=10, n=4) | 70.40 [59.41 to 81.39] | 47.00 [42.50 to 51.50] | 58.25 [41.24 to 75.26]
  Day 7 (20 μM ADP) (n=5, n=10, n=5) | 71.00 [53.46 to 88.54] | 58.30 [53.14 to 63.46] | 73.20 [55.55 to 90.85]
  Day 9 (20 μM ADP) (n=5, n=10, n=5) | 62.40 [41.97 to 82.83] | 62.00 [52.20 to 71.80] | 68.60 [59.44 to 77.76]
  Day 11 (20 μM ADP) (n=5, n=10, n=5) | 72.00 [59.59 to 84.41] | 65.20 [58.11 to 72.29] | 63.80 [33.21 to 94.39]
  Baseline (5 μM ADP) (n=5, n=10, n=6) | 64.40 [60.21 to 68.59] | 62.60 [55.76 to 69.44] | 70.67 [65.42 to 75.91]
  Day 1 (5 μM ADP) (n=5, n=10, n=6) | 39.40 [23.40 to 55.40] | 22.00 [15.37 to 28.63] | 25.50 [18.18 to 32.82]
  Day 3 (5 μM ADP) (n=5, n=10, n=6) | 50.20 [36.31 to 64.09] | 32.80 [28.73 to 36.87] | 48.67 [38.85 to 58.48]
  Day 5 (5 μM ADP) (n=5, n=10, n=4) | 64.20 [48.17 to 80.23] | 39.50 [34.26 to 44.74] | 53.25 [38.23 to 68.27]
  Day 7 (5 μM ADP) (n=5, n=10, n=5) | 60.40 [40.90 to 79.90] | 52.40 [44.95 to 59.85] | 65.40 [46.91 to 83.89]
  Day 9 (5 μM ADP) (n=5, n=10, n=5) | 58.40 [35.53 to 81.27] | 56.00 [46.46 to 65.54] | 60.00 [51.55 to 68.45]
  Day 11 (5 μM ADP) (n=5, n=10, n=5) | 61.80 [50.53 to 73.07] | 58.90 [51.85 to 65.95] | 56.00 [29.54 to 82.46]

10. Secondary Outcome: Extent of Initial Inhibition of Platelet Aggregation to the Return of Baseline Platelet Function: Multiplate® ADP Test and ADP Test High Sensitivity (HS)
Description: Return of baseline platelet function was assessed by Multiplate® ADP test and ADP test High Sensitivity (HS). Multiplate analyzer was used to assess platelet aggregation based on impedance aggregometry in whole blood. The agonist ADP was added to stirred whole blood after dilution (1:2 with 0.9% NaCl solution) in a final concentration of 6.4 µM (ADP Test) or in final concentration of 6.4 µM ADP plus 9.4 nM Prostaglandin E1 (PGE1) (ADPtest HS). Platelet aggregation was continuously recorded for 5 minutes and quantified as area under the aggregation curve (AUC=AU*min) of aggregation units (AU).
Time Frame: Up through 11 days
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: Aggregation Units * minutes
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 5 | 10 | 6
Aggregation Units * minutes
  Baseline (ADP) (n=5, n=10, n=6) | 536.60 [453.01 to 620.19] | 601.60 [489.12 to 714.08] | 459.33 [369.59 to 549.07]
  Day 1 (ADP) (n=5, n=10, n=6) | 248.80 [133.88 to 363.72] | 90.00 [74.08 to 105.92] | 118.17 [79.82 to 156.51]
  Day 3 (ADP) (n=5, n=10, n=6) | 347.60 [97.50 to 597.70] | 140.90 [96.21 to 185.59] | 134.67 [100.88 to 168.46]
  Day 5 (ADP) (n=5, n=10, n=4) | 428.40 [265.81 to 590.99] | 231.30 [173.02 to 289.58] | 296.00 [164.77 to 427.23]
  Day 7 (ADP) (n=5, n=10, n=5) | 478.80 [338.41 to 619.19] | 316.20 [257.51 to 374.89] | 295.40 [229.77 to 361.03]
  Day 9 (ADP) (n=5, n=10, n=5) | 529.40 [381.37 to 677.43] | 549.00 [439.70 to 658.30] | 484.40 [316.20 to 652.60]
  Day 11 (ADP) (n=5, n=10, n=5) | 555.00 [431.41 to 678.59] | 500.20 [426.84 to 573.56] | 564.00 [439.67 to 688.33]
  Baseline (ADP HS) (n=5, n=10, n=6) | 361.00 [225.47 to 496.53] | 411.70 [330.83 to 492.57] | 344.00 [246.05 to 441.95]
  Day 1 (ADP HS) (n=5, n=10, n=6) | 166.80 [88.39 to 245.21] | 34.50 [18.08 to 50.92] | 70.17 [40.54 to 99.80]
  Day 3 (ADP HS) (n=5, n=10, n=6) | 257.60 [41.96 to 473.24] | 79.30 [55.45 to 103.15] | 90.50 [64.84 to 116.16]
  Day 5 (ADP HS) (n=5, n=10, n=4) | 256.80 [118.58 to 395.02] | 114.10 [87.86 to 140.34] | 145.00 [72.29 to 217.71]
  Day 7 (ADP HS) (n=5, n=10, n=5) | 263.60 [124.99 to 402.21] | 189.50 [152.93 to 226.07] | 170.60 [115.78 to 225.42]
  Day 9 (ADP HS) (n=5, n=10, n=5) | 388.20 [172.68 to 603.72] | 344.60 [263.97 to 425.23] | 343.60 [228.01 to 459.19]
  Day 11 (ADP HS) (n=5, n=10, n=5) | 373.20 [256.35 to 490.05] | 365.40 [294.25 to 436.55] | 404.00 [329.60 to 478.40]

11. Secondary Outcome: Mean Number of Days to the Return of Baseline Platelet Function in All Treatment Arms (Adjusted for Level of Inhibition 24 Hours Post-LD) by LTA (5 and 20 μM ADP)
Description: Maximum platelet aggregation (MPA) to 5 and 20 μM ADP were assessed by LTA. This outcome measure was not analyzed due to limited sample size.
Time Frame: Up through 11 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Mean Number of Days to the Return of Baseline Platelet Function in All Treatment Arms (Adjusted for Level of Inhibition 24 Hrs Post-LD) by Multiplate® ADP Test and ADP Test High Sensitivity (HS)
Description: The Multiplate analyzer was used to assess platelet aggregation based on impedance aggregometry in whole blood. After adding 6.4 µM ADP (ADP test) or 6.4 µM ADP plus 9.4 nM Prostaglandin E1 (PGE1) (ADP test HS), area under the aggregation curve (AUC) was calculated. This outcome measure was not analyzed due to limited sample size.
Time Frame: Up through 11 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Platelet Function by LTA at 5 and 20 μM ADP
Description: MPA to 5 and 20 μM ADP were assessed by LTA.
Time Frame: 24 hours post-loading dose
Population: LD ITT population: All randomized participants who received an LD with evaluable PD measurements 24 hours post-LD.
Measure: Mean (Standard Deviation); unit: percent aggregation
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 5 | 10 | 6
percent aggregation
  Maximum Aggregation (20 µM ADP) | 52.60 (20.60) | 27.30 (10.86) | 31.67 (11.13)
  Maximum Aggregation (5 µM ADP) | 39.40 (16.79) | 22.00 (11.44) | 25.50 (8.89)

14. Secondary Outcome: Platelet Function by Multiplate® ADP Test and ADP Test HS
Description: The Multiplate analyzer was used to assess platelet aggregation based on impedance aggregometry in whole blood. After adding 6.4 µM ADP (ADP test) or 6.4 µM ADP plus 9.4 nM PGE1 (ADP test HS), area under the aggregation curve (AUC) were calculated.
Time Frame: 24 hours post-loading dose
Population: LD ITT Population: All randomized participants who received an LD with evaluable PD measurements 24 hours post-LD.
Measure: Mean (Standard Deviation); unit: aggregation units*minute
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Number analyzed (Participants) | 5 | 10 | 6
aggregation units*minute
  ADP Test AUC | 248.80 (120.54) | 90.00 (27.46) | 118.17 (46.61)
  ADP Test HS AUC | 166.80 (82.24) | 34.50 (28.33) | 70.17 (36.02)

ADVERSE EVENTS:
Arm/Group | Clopidogrel 600 mg | Prasugrel 60 mg | Prasugrel 30 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel 600 mg (N=10) | Prasugrel 60 mg (N=10) | Prasugrel 30 mg (N=8)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial was terminated early due to enrollment futility which resulted in limited data and the inability to analyze some outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days